CLINICAL TRIAL: NCT00176462
Title: CINJALL: Treatment for Children With Acute Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 020101; 0220003389 (Other: IRB Number); P30CA072720 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-05

CONDITIONS: Acute Lymphocytic Leukemia
Keywords: Acute Lymphocytic Leukemia; Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — Aminopterin; Asparaginase; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Mercaptopurine; Methotrexate; Thioguanine; Vincristine; Hydrocortisone; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 Standard Risk (Experimental): 6-MERCAPTOPURINE DAUNOMYCIN DEXAMETHASONE Triple Intrathecal Therapy (ITT) L-ASPARAGINASE VINCRISTINE METHOTREXATE Leucovorin
  Interventions: Drug: L-asparaginase; Drug: daunomycin; Drug: dexamethasone; Drug: 6-mercaptopurine; Drug: methotrexate; Drug: vincristine; Drug: Triple Intrathecal Therapy (MTX, Cytarabine, Hydrocortisone); Drug: Leucovorin
- Arm 2 High Risk (Experimental): 6-MERCAPTOPURINE DAUNOMYCIN DEXAMETHASONE Triple Intrathecal Therapy (ITT) L-ASPARAGINASE VINCRISTINE 6-THIOGUANINE CYTARABINE AMINOPTERIN CYCLOPHOSPHAMIDE ARABINOSIDE-C
  Interventions: Drug: aminopterin; Drug: L-asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunomycin; Drug: dexamethasone; Drug: 6-mercaptopurine; Drug: 6-thioguanine; Drug: vincristine; Drug: Triple Intrathecal Therapy (MTX, Cytarabine, Hydrocortisone); Drug: Leucovorin

INTERVENTIONS:
Drug: aminopterin — Therapy will be divided into five phases: Induction, Consolidation, Delayed Intensification (only for those patients meeting clinical criteria defining a high risk of relapse), Intensive Continuation, and Continuation
  Arms: Arm 2 High Risk
Drug: L-asparaginase — Therapy will be divided into five phases: Induction, Consolidation, Delayed Intensification (only for those patients meeting clinical criteria defining a high risk of relapse), Intensive Continuation, and Continuation
Drug: cyclophosphamide — Therapy will be divided into five phases: Induction, Consolidation, Delayed Intensification (only for those patients meeting clinical criteria defining a high risk of relapse), Intensive Continuation, and Continuation
  Arms: Arm 2 High Risk
Drug: cytarabine — Therapy will be divided into five phases: Induction, Consolidation, Delayed Intensification (only for those patients meeting clinical criteria defining a high risk of relapse), Intensive Continuation, and Continuation
  Arms: Arm 2 High Risk
Drug: daunomycin — Therapy will be divided into five phases: Induction, Consolidation, Delayed Intensification (only for those patients meeting clinical criteria defining a high risk of relapse), Intensive Continuation, and Continuation
Drug: dexamethasone — Therapy will be divided into five phases: Induction, Consolidation, Delayed Intensification (only for those patients meeting clinical criteria defining a high risk of relapse), Intensive Continuation, and Continuation
Drug: 6-mercaptopurine — Therapy will be divided into five phases: Induction, Consolidation, Delayed Intensification (only for those patients meeting clinical criteria defining a high risk of relapse), Intensive Continuation, and Continuation
Drug: methotrexate — Therapy will be divided into five phases: Induction, Consolidation, Delayed Intensification (only for those patients meeting clinical criteria defining a high risk of relapse), Intensive Continuation, and Continuation
  Arms: Arm 1 Standard Risk
Drug: 6-thioguanine — Therapy will be divided into five phases: Induction, Consolidation, Delayed Intensification (only for those patients meeting clinical criteria defining a high risk of relapse), Intensive Continuation, and Continuation
  Arms: Arm 2 High Risk
Drug: vincristine — Therapy will be divided into five phases: Induction, Consolidation, Delayed Intensification (only for those patients meeting clinical criteria defining a high risk of relapse), Intensive Continuation, and Continuation
Drug: Triple Intrathecal Therapy (MTX, Cytarabine, Hydrocortisone)
Drug: Leucovorin

SUMMARY:
The purpose of this research study is to identify better ways to treat children and young adults with acute lymphocytic leukemia (ALL). At the same time, doctors hope to define methods to identify those patients at higher risk for certain side effects, as well as those who are at higher risk for relapse of their leukemia.

DETAILED DESCRIPTION:
Outline of Therapy:

Combinations of chemotherapy drugs will be given orally, intravenously and intrathecally (directly into the cerebrospinal fluid by spinal tap) over a period of roughly two and a half years.

Therapy will be divided into five phases:

Induction (4 weeks): chemotherapy given to produce a clinical remission (defined by normal blood counts, with the absence of leukemia cells in the blood and fewer than 5% leukemia cells in the bone marrow).

Consolidation (11 weeks): chemotherapy given to consolidate the remission. Delayed Intensification (7 weeks) Intensive chemotherapy aimed at killing any resistant leukemia cells will be given only for patients at high risk of relapse.

Intensive Continuation (approximately 1 year): Eight week cycles of chemotherapy, given eight times.

Continuation (final year of therapy): Eight week cycles of largely oral chemotherapy, with one clinic visit for a lumbar puncture every eight weeks.

Irradiation: radiation will be given in the middle of intensive continuation to the head and spine of those patients who have leukemia cells found in the cerebrospinal fluid at the time of diagnosis.

Follow-up: After the conclusion of therapy, there will be periodic office visits, initially monthly, then gradually spaced out to annual visits. The purpose of these visits is to evaluate for late side-effects of therapy.

ELIGIBILITY:
Inclusion:

* Newly Diagnosed ALL, excluding mature B-cell ALL (surface Ig positive)
* Patients with overt CNS (central nervous system) or testicular disease are eligible
* Informed consent according to institutional and FDA guidelines.
* Adequate organ function is required.
* HIV seropositive patients will not be excluded from this study.
* Patients greater than 1 year of age and less than 29.99 years of age are eligible.

Exclusion Criteria

* Patients with medical, psychological, or psychiatric problems that are likely to compromise their ability to tolerate intensive therapy will be ineligible.
* All patients with evidence of significant organ dysfunction not thought to be attributable to ALL (patients with clinically significant congestive heart failure, cardiac ejection fraction <40%, total bilirubin >2, serum creatinine >2) will be ineligible. Note: echocardiogram or MUGA are required prior to therapy ONLY for those patients with history or physical findings suggestive of cardiac dysfunction not directly attributable to anemia or ALL. Note: Patients with total bilirubin >2 but direct (conjugated) bilirubin less than the upper limit of normal will still be eligible. These patients should be evaluated for deficiency of the enzyme glucuronyl transferase.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2001-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barton Kamen, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (2):
- United States (2):
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 59 patients with ALL were enrolled between March, 2001 and September, 2005 at the Cancer Institute of New Jersey (outpatient clinical research facility) and 1 patient was enrolled at Jersey Shore University Medical Center (a community hospital).
Period: Induction (4 Weeks)
Arm/Group | Arm 1 Standard Risk | Arm 2 High Risk
Started | 21 | 39
Completed | 20 | 34
Not Completed | 1 | 5
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Death | 1 | 2
Not completed — Lack of Efficacy | 0 | 1
Period: Consolidation (12 Weeks)
Arm/Group | Arm 1 Standard Risk | Arm 2 High Risk
Started | 20 | 34
Completed | 20 | 29
Not Completed | 0 | 5
Not completed — Patient moved to another state | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 0 | 2
Not completed — Not documented | 0 | 1
Period: Delayed Intensification (8 Weeks)
Arm/Group | Arm 1 Standard Risk | Arm 2 High Risk
Started | 20 | 29
Completed | 20 | 29
Not Completed | 0 | 0
Period: Intensive Continuation (8X8-week Cycles)
Arm/Group | Arm 1 Standard Risk | Arm 2 High Risk
Started | 20 | 29
Completed | 19 | 26
Not Completed | 1 | 3
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 0 | 3
Period: Continuation -up to 30mos Post Remission
Arm/Group | Arm 1 Standard Risk | Arm 2 High Risk
Started | 19 | 26
Completed | 19 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 Standard Risk | Arm 2 High Risk | Total
Number analyzed (Participants) | 21 | 39 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21 | 30 | 51
  Between 18 and 65 years | 0 | 9 | 9
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.71 (1.77) | 16 (9.8) | 11.7 (9.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 18 | 29
  Male | 10 | 21 | 31
Region of Enrollment [Number; unit: participants]
  United States | 21 | 39 | 60

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With ALL at High Risk of Relapse (Arm 2) Who Were Relapse-free at 5 Years
Description: This measure looks at the percentage of patients on Arm 2 who did not experience a relapse at 5 years, where relapse is defined as the presence of progressive disease after the achievement of a complete remission.
Time Frame: 5 years
Population: Number of high risk ALL patients treated.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 2 High Risk
Number analyzed (Participants) | 37
percentage of participants | 64.9

2. Secondary Outcome: To Measure 5-methyltetrahydrofolate, Aminopterin and Methotrexate Uptake in Leukemic Blasts Isolated at Diagnosis
Time Frame: 5 years
Population: We did not analyze this outcome measure. The laboratory analysis was not performed. The Principal Investigator left the institution.
Arm/Group | Arm 1 Standard Risk | Arm 2 High Risk
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 7 years, 6 months
Arm/Group | Arm 1 Standard Risk | Arm 2 High Risk
Serious Adverse Events (participants affected / at risk) | 20/21 | 36/39
Other Adverse Events (participants affected / at risk) | 21/21 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 Standard Risk (N=21) | Arm 2 High Risk (N=39)
Platelets (Blood and lymphatic system disorders) | 5 (5) | 5 (7)
Thrombosis/embolism (General disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 1 (1) | 1 (2) — in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L
Febrile neutropenia (Infections and infestations) | 16 (29) | 17 (35)
Infection with unknown ANC (Infections and infestations) | 1 (1) | 3 (3)
Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (Infections and infestations) | 1 (1) | 2 (2)
Infection without neutropenia (Infections and infestations) | 3 (3) | 1 (1)
Neurology (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Neuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Allergic reaction/hypersensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (7)
Dehydration (Gastrointestinal disorders) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain or cramping (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis / pharyngitis (Gastrointestinal disorders) | 0 (0) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Anorexia (General disorders) | 0 (0) | 3 (3)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypokalemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 3 (4)
Fibrinogen (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
DIC (disseminated intravascular coagulation) (Vascular disorders) | 0 (0) | 2 (2)
Typhlitis (inflammation of cecum) (Gastrointestinal disorders) | 0 (0) | 2 (2)
Psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Leukocytes (total WBC) - Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4)
Fatigue (General disorders) | 0 (0) | 1 (1)
Broncohspasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperglycemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Neuropathic pain (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Syncope (General disorders) | 0 (0) | 2 (2)
Melena/GI bleeding - Hemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac troponin I (Cardiac disorders) | 0 (0) | 1 (1)
Relapsed leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 Standard Risk (N=21) | Arm 2 High Risk (N=39)
Platelets (Blood and lymphatic system disorders) | 1 (1) | 3 (4)
Fever (General disorders) | 12 (22) | 15 (21)
Infection with unknown ANC (Infections and infestations) | 1 (1) | 4 (4)
Infection without neutropenia (Infections and infestations) | 1 (1) | 1 (1)
Neuropathy (Nervous system disorders) | 0 (0) | 3 (3)
Allergic reaction/hypersensitivity (Immune system disorders) | 3 (4) | 0 (0)
Dehydration (Gastrointestinal disorders) | 1 (1) | 5 (6)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (9)
Vomiting (Gastrointestinal disorders) | 2 (2) | 7 (17)
Headache - Pain-Head (General disorders) | 0 (0) | 7 (10)
Speech impairment (Nervous system disorders) | 0 (0) | 1 (3)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain or cramping (Gastrointestinal disorders) | 1 (1) | 4 (4)
Stomatitis / pharyngitis (Gastrointestinal disorders) | 1 (1) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Appendicitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Other Toxicity (General disorders) | 3 (3) | 5 (5)
Otitis middle ear (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Extremity pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 2 (2)
Muscle Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Vascular disorders) | 0 (0) | 1 (1)
Hypokalemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Seizure(s) (Nervous system disorders) | 0 (0) | 1 (2)
Weight gain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Edema (Pulmonary) (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rigors (General disorders) | 0 (0) | 1 (2)
Neurology - Mood Alteration (Nervous system disorders) | 0 (0) | 1 (1)
GI other (Elevated liver enzymes) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hyperammonemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Excessive thirst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyperglycemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Urinary freqency (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypercalcemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrythmia (Cardiac disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Infection / Febrile neutropenia (Infections and infestations) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 1 (1)
Ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Phlebitis (superficial) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Amylase (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fever & pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Antifolate therapy was non-randomly assigned, therefore, we do not have a statistical basis to compare the toxicity observed among patients on the standard risk and high risk treatment arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes